CLINICAL TRIAL: NCT01182493
Title: OpT2mise Glucose Control in Type 2 DM With Insulin Pump Therapy
Brief Title: OpT2mise Glucose Control in Type 2 Diabetes Mellitus (DM) With Insulin Pump Therapy
Acronym: OpT2mise
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Medtronic Diabetes (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: EUR05 / CEP234
Record Dates: First submitted 2010-08-11; First posted 2010-08-16 (Estimated); Results first posted 2016-03-15 (Estimated); Last update posted 2018-03-12 (Actual); Status verified 2018-02

CONDITIONS: Diabetes Mellitus, Type 2
Keywords: Diabetes Mellitus; MDI; pump therapy
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Diabetes Mellitus

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Insulin Pump Treatment (Experimental): Patients will get an insulin pump
  Interventions: Device: Insulin Pump (Medtronic Minimed Paradigm® VEO)
- Insulin treatment with MDI (No Intervention): patients treated with Multiple Daily Injections (MDI); basal/bolus therapy with rapid- and long-acting analogs with at least 3 injections per day

INTERVENTIONS:
Device: Insulin Pump (Medtronic Minimed Paradigm® VEO) — The pump delivers insulin as specified by the patient
  Other Names: Medtronic MiniMed Paradigm® VEO system (MMT-554/754
  Arms: Insulin Pump Treatment

SUMMARY:
The purpose of this study is to evaluate the comparative effectiveness of insulin pump therapy versus multiple daily injections in insulin-taking type 2 Diabetes Mellitus who are sub optimally controlled with multiple daily injections (MDI).

DETAILED DESCRIPTION:
The type of study is interventional post-market release. All the devices under investigation have CE mark, and are used within intended use.

This study has been designed to be prospective randomized controlled with a single-arm cross-over in the continuation phase.

Four hundred type 2 Multiple Daily Injections (MDI) treated patients will undergo a screening (run-in) phase of 8 weeks. The aim of the screening phase is to eliminate the study effect that might result in a decrease of HbA1c and to make sure that patients, who are failing current MDI therapy, are selected.

After this screening phase, eligible patients will be randomised to receive either Continuous Subcutaneous Insulin Infusion (CSII) treatment or continue MDI treatment. The study phase is a 6-months phase with 2-arms parallel design.

ELIGIBILITY:
Inclusion Criteria at screening:

1. Diagnosed with type 2 DM, as per Investigator discretion
2. HbA1c (DCCT-standard) must be ≥ 8.0% and ≤12% as evidenced by central lab value taken at screening
3. Insulin resistance defined as required daily dose between 0.5-1.8 U/Kg or a maximum of 220 units of insulin per day
4. Aged 30 to 75 years old (inclusive)
5. On MDI regimen (basal/bolus regimen with long-acting insulin and rapid acting analogs) defined as ≥ 3 injections per day for at least 3 months prior signing the informed consent
6. Ability to comply with technology, according to Investigator's judgment
7. Patients must be willing to undergo all study procedures
8. Female patients of child-bearing potential must be using adequate contraception means as assessed by Investigator

at randomisation:

1. Diagnosed with type 2 DM, as per Investigator discretion
2. HbA1c (DCCT-standard) must be ≥ 8.0% and ≤12% as evidenced by central lab value
3. Insulin resistance defined as required daily dose between 0.7-1.8 U/Kg or a maximum of 220 units of insulin per day
4. On MDI (basal/bolus regimen with long-acting insulin and rapid acting analogs) defined as ≥ 3 injections per day
5. Ability to comply with technology, according to Investigator's judgment
6. ≥ 2.5 SMBG per day on average, as reported in Carelink clinical during the run-in phase.
7. Patients must be willing to undergo all study procedures
8. Female patients of child-bearing potential must be using adequate contraception means as assessed by Investigator

Exclusion Criteria :

1. Subject has a history (≥ 2 events) of hypoglycemic seizure or hypoglycemic coma within the last 6 months
2. Subject is pregnant as assessed by a pregnancy test with central laboratory, or plans to become pregnant during the course of the study
3. Participation in another interventional clinical study, on-going or completed less than 3 months prior to signature of Patient Informed Consent.
4. Subject has proliferative retinopathy or sight threatening maculopathy
5. Subject has

   * an acute coronary syndrome (myocardial infarction or unstable angina) within 12 months OR
   * coronary artery revascularization by bypass surgery or stenting within 3 months OR
   * a transient ischemic attack (TIA) or cerebrovascular accident (CVA) within 3 months OR
   * hospitalization for heart failure within 3 months or current New York Functional Class III or IV OR
   * current 2nd or 3rd degree heart block OR
   * symptomatic ventricular rhythm disturbances OR
   * thromboembolic disease within the last 3 months OR
   * 2nd degree Mobitz type II or 3rd degree heart block
6. Subject with renal impairment expressed as estimated glomerular filtration rate (eGFR) using the Modification of Diet in Renal Disease (MDRD) formula < 30 ml/min as demonstrated by the screening central laboratory value at the time of enrollment
7. Subject has taken oral or injectable steroids within the last 30 days
8. Systolic blood pressure on screening visit is > 180 mmHg
9. Diastolic blood pressure on screening visit is > 110 mmHg
10. Any other disease (eg active cancer under treatment) or condition including abnormalities found on the screening tests, that in the opinion of the Investigator, may preclude him/her from participating in the study
11. Taking any medication prescribed for weight loss
12. Alcohol or drug abuse, other than nicotine, at the investigator's discretion
13. Use of a GLP-1 agonist or pramlintide (Symlin)

Ages: 30 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 331 (Actual)
Dates: Start 2010-12; Primary Completion 2014-02 (Actual); Study Completion 2014-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ohad Cohen, MD, Principal Investigator — Chaim Sheba Medical Center, Tel Hashomer, Israel; Ignacio Conget, MD, Principal Investigator — ICMDM Hospital Clínic i, Barcelona, Spain; Yves Reznic, MD, Principal Investigator — CHU Côte de Nacre, France; Ronnie Aronson, MD, Principal Investigator — FRCPC, FACE LMC Endocrinology Centres, Canada
Locations (36):
- United States (3):
  - Atlanta Diabetes Associates, Atlanta, Georgia
  - Albany Medical College, Albany, New York
  - SUNY Upstate Medical University, Syracuse, New York
- City hopital Vienna-Hieting, Vienna, Austria
- Canada (8):
  - Clinical Professor Department of Medicine University of Calgary, Calgary, Alberta
  - Endocrinologist, 202-301 Columbia Street East, New Westminster, British Columbia
  - 416-1033 Davie St, Vancouver, British Columbia
  - Health Science Centre, St. John's, Newfoundland and Labrador
  - LMC Endocrinology Centre, Oakville, Ontario
  - Canadian Centre for Research on Diabetes, Smiths Falls, Ontario
  - Toronto General Hsopital, Toronto, Ontario
  - McGill University, McGill Nutrition and Food Science Centre, Montreal, Quebec
- France (6):
  - CHU Côte de Nacre, Caen
  - CHU - Ste Marguerite, Marseille
  - Hopital Lapeyronie, Montpellier
  - CHU de Nancy, Nancy
  - CHU Strasbourg, Strasbourg
  - CHU Toulouse Rangueil, Toulouse
- Germany (2):
  - Fachklinik Bad Heilbrunn, Bad Heilbrunn
  - Zentrum für Diabetes und Gefäßerkrankungen, Münster
- Péterfy Hospital and Emergency Center Diabetes Outpatient Clinic, Budapest, Hungary
- Israel (4):
  - Soroka University Medical Center, Beersheba
  - Diabetic Clinic, Jerusalem
  - Chaim Sheba Medical center Endocrinology unit, Tel Hashomer - Ramat Gan
  - Assaf- Harofeh Medical Center, Ẕerifin
- Italy (3):
  - Università degli Studi di Bari - Policlinico Universitario, Bari
  - Universita di Perugia - Ospedale S.M. Della Misericordia, Perugia
  - University La Sapienza - Policlinico, Roma
- Netherlands (3):
  - IJsselland Ziekenhuis Poli Interne geneeskunde, Capelle aan den IJssel
  - Maxima Medisch Centrum, Eindhoven
  - Bethesda Diabetes Research Center, Hoogeveen
- University Clinic of Endocrinology, Skopje, North Macedonia
- Clinic for Endocrinology, Diabetes and Metabolic Diseases, Belgrade, Serbia
- South Africa (2):
  - Centre for Diabetes and Endocrinology, Johannesburg
  - Dr.Garcjan Podgorski, Port Elizabeth
- ICMDM Hospital Clínic i Universitari, Barcelona, Spain

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Chlup R, Runzis S, Castaneda J, Lee SW, Nguyen X, Cohen O. Complex Assessment of Metabolic Effectiveness of Insulin Pump Therapy in Patients with Type 2 Diabetes Beyond HbA1c Reduction. Diabetes Technol Ther. 2018 Feb;20(2):153-159. doi: 10.1089/dia.2017.0283. Epub 2017 Dec 7. PMID 29215299
- [Derived] Metzger M, Castaneda J, Reznik Y, Giorgino F, Conget I, Aronson R, de Portu S, Runzis S, Lee SW, Cohen O. Factors associated with improved glycemic control following continuous subcutaneous insulin infusion therapy in patients with type 2 diabetes uncontrolled with bolus-basal insulin regimens: An analysis from the OpT2mise randomized trial. Diabetes Obes Metab. 2017 Oct;19(10):1490-1494. doi: 10.1111/dom.12960. Epub 2017 Jul 25. PMID 28374511
- [Derived] Reznik Y, Cohen O, Aronson R, Conget I, Runzis S, Castaneda J, Lee SW; OpT2mise Study Group. Insulin pump treatment compared with multiple daily injections for treatment of type 2 diabetes (OpT2mise): a randomised open-label controlled trial. Lancet. 2014 Oct 4;384(9950):1265-72. doi: 10.1016/S0140-6736(14)61037-0. Epub 2014 Jul 2. PMID 24998009

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 36 hospitals, tertiary care centres, and referal centres participated: eight in Canada, 23 in Europe and Israel, two in South Africa, and three in the USA. The study started in December 2010, and the fi nal data collection date for the primary outcome measure was in February 2014
Period: Overall Study
Arm/Group | Insulin Pump Treatment | Insulin Treatment With MDI
Started | 168 | 163
Completed | 152 | 156
Not Completed | 16 | 7

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Insulin Pump Treatment | Insulin Treatment With MDI | Total
Number analyzed (Participants) | 168 | 163 | 331
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 168 | 163 | 331
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 55.5 (9.7) | 56.4 (9.5) | 56.0 (9.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 74 | 77 | 151
  Male | 94 | 86 | 180
HbA1c [Mean (Standard Deviation); unit: % of glycosylated hemoglobin] | 9.0 (0.75) | 9.0 (0.76) | 9.0 (0.75)

OUTCOME MEASURES:

1. Primary Outcome: Between Group Difference in HbA1c When Comparing CSII to MDI
Description: To evaluate change in glycemic control (HbA1c) after 6 months of insulin pump therapy in patients with type 2 DM, as compared to patients on MDI therapy over the same time period. Change in A1c = A1c at 6 month - A1c at baseline
Time Frame: baseline and 6 months
Measure: Mean (Standard Deviation); unit: Change in % HbA1c
Arm/Group | Insulin Pump Treatment | Insulin Treatment With MDI
Number analyzed (Participants) | 168 | 163
Change in % HbA1c | -1.1 (1.2) | -0.4 (1.1)

2. Secondary Outcome: Change in Glycemic Variability - AUC in Hypo (≤70mg/dL)
Description: Glycemic parameters calculated from blinded CGM data: change in AUC (Area Under the Curve) in hypo- (≤70mg/dL), among subjects with available AUC results. Change in hypo AUC = hypo AUC at 6 month - hypo AUC at baseline
Time Frame: 6 months
Measure: Mean (Standard Deviation); unit: mg/dL/min
Arm/Group | Insulin Pump Treatment | Insulin Treatment With MDI
Number analyzed (Participants) | 113 | 108
mg/dL/min | 0 (0.6) | -0.1 (0.9)

3. Secondary Outcome: Safety - Severe Hypoglycemia Incidence
Description: Severe hypoglycemia incidence during the study
Time Frame: 6 months
Measure: Count of Participants; unit: Participants
Arm/Group | Insulin Pump Treatment | Insulin Treatment With MDI
Number analyzed (Participants) | 168 | 163
Participants | 0 | 1

4. Secondary Outcome: Change in Glycemic Variability - AUC in Hyper (≥180mg/dL)
Description: Glycemic parameters calculated from blinded CGM data: change in AUC (Area Under the Curve) in hyper- (≥180mg/dL), among subjects with available AUC results. Change in hyper AUC = hyper AUC at 6 month - hyper AUC at baseline
Time Frame: 6 months
Measure: Mean (Standard Deviation); unit: mg/dL/min
Arm/Group | Insulin Pump Treatment | Insulin Treatment With MDI
Number analyzed (Participants) | 113 | 108
mg/dL/min | -11 (26.3) | -2.6 (17.4)

5. Secondary Outcome: Quality of Life and Treatment Satisfaction - Results From Diabetes Treatment Satisfaction Questionnaire (DTSQ)
Description: Subjects were asked to complete the Diabetes Treatment Satisfaction Questionnaire (DTSQs). Treatment satisfaction is measured by means of the DTSQs, status version (DTSQs, Bradley, 1990). It consists of a six-item scale assessing treatment satisfaction (TS) and two items assessing perceived frequency of hyperglycaemia and hypoglycaemia. The DTSQs items are scored on a scale from 0 to 6. The scale total is computed by adding the six items 1, 4, 5, 6, 7, and 8, to produce the Treatment Satisfaction scale total, which has a min of 0 and a max of 36. Higher score at 6 month compared to baseline represents a better outcome. Change in treatment satisfaction = score at 6 month - score at baseline, among subjects with available satisfaction scores
Time Frame: 6 months
Measure: Mean (Standard Deviation); unit: score
Arm/Group | Insulin Pump Treatment | Insulin Treatment With MDI
Number analyzed (Participants) | 140 | 143
score | 4.75 (6.9) | -0.26 (6.9)

6. Secondary Outcome: Change in Body Weight
Description: Change in body weight from randomization to the end of study. Change in body weight = weight at 6 month - weight at baseline, among subjects with available body weight
Time Frame: 6 months
Measure: Mean (Standard Deviation); unit: kg
Arm/Group | Insulin Pump Treatment | Insulin Treatment With MDI
Number analyzed (Participants) | 151 | 154
kg | 1.52 (3.53) | 1.12 (3.62)

7. Secondary Outcome: Safety - Diabetic Ketoacidosis Incidence
Description: Diabetic Ketoacidosis incidence during the study
Time Frame: 6 Months
Measure: Count of Participants; unit: Participants
Arm/Group | Insulin Pump Treatment | Insulin Treatment With MDI
Number analyzed (Participants) | 168 | 163
Participants | 0 | 0

ADVERSE EVENTS:
Time Frame: All adverse events reported during the study period (6 months)
Arm/Group | Insulin Pump Treatment | Insulin Treatment With MDI
All-Cause Mortality (participants affected / at risk) | 0/168 | 0/163
Serious Adverse Events (participants affected / at risk) | 13/168 | 10/163
Other Adverse Events (participants affected / at risk) | 108/168 | 99/163
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Insulin Pump Treatment (N=168) | Insulin Treatment With MDI (N=163)
Cellulitis on left lower abdomen (Infections and infestations) | 1 (1) | 0 (0)
Exacerbation of Hypertension (Vascular disorders) | 1 (1) | 0 (0)
Retinal Hemorrhage Right Eye (Eye disorders) | 1 (1) | 0 (0)
acute coronary syndrome (Cardiac disorders) | 1 (1) | 0 (0)
Endometrial Cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
abscess (Infections and infestations) | 1 (1) | 0 (0)
chronic hyperglycemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
tachycardia (Cardiac disorders) | 1 (1) | 0 (0)
CARDIAC ARYTHMIA WITH ATRIAL FIBRILLATION (Cardiac disorders) | 1 (1) | 0 (0)
chest pain (General disorders) | 1 (1) | 0 (0)
coronary artery bypass graft (Surgical and medical procedures) | 1 (1) | 0 (0)
PNEUMONIA (Infections and infestations) | 1 (1) | 0 (0)
acute pancreatitis (Gastrointestinal disorders) | 1 (1) | 0 (0)
postmenopausal bleeding with abnormality of cervix, hyperplasia (Reproductive system and breast disorders) | 1 (1) | 0 (0)
Congestive Heart Failure (Cardiac disorders) | 1 (1) | 0 (0)
Knee arthrosis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Ketosis (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Spinal stenosis L1-L2 (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Hepatic abscess (Infections and infestations) | 0 (0) | 1 (1)
Worsening Hepatic Abscess (Infections and infestations) | 0 (0) | 1 (1)
Pancreatitis (Gastrointestinal disorders) | 0 (0) | 1 (1)
heart Failure (Cardiac disorders) | 0 (0) | 1 (1)
abdominal pain (Gastrointestinal disorders) | 0 (0) | 1 (1)
hyperglycemia with ketosis without acidosis (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Hepatic Encephalophthy (Nervous system disorders) | 0 (0) | 1 (1)
Atypical Ductal Hyperplasia (General disorders) | 0 (0) | 1 (1)
Hepatocellular carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Chest Pain (non cardiac) (General disorders) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Insulin Pump Treatment (N=168) | Insulin Treatment With MDI (N=163)
ANEMIA (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
SWOLLEN LYMPH NODES (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
ATRIAL FIBRILLATION REOCCURENCE (Cardiac disorders) | 1 (1) | 0 (0)
CARDIAC INSUFFICIENCY (Cardiac disorders) | 0 (0) | 1 (1)
CONGESTIVE HEART FAILURE (Cardiac disorders) | 1 (1) | 0 (0)
HEART BEATING PALPITATIONS (Cardiac disorders) | 0 (0) | 1 (1)
ISCHEMIC CARDIOMYOPATHY (Cardiac disorders) | 0 (0) | 1 (1)
MIOCARDIAL INFARCTION (Cardiac disorders) | 0 (0) | 1 (1)
MITRAL INSUFFICIENCY (Cardiac disorders) | 0 (0) | 1 (1)
PALPITATIONS (Cardiac disorders) | 0 (0) | 1 (1)
SINUSTACHYCARDIA (Cardiac disorders) | 1 (1) | 1 (1)
BLOCKED RIGHT EAR (Ear and labyrinth disorders) | 1 (1) | 0 (0)
HEARING LOSS (Ear and labyrinth disorders) | 1 (1) | 0 (0)
PERICHONDRITIS OF HUMEROSCAPULAR JOINT (Ear and labyrinth disorders) | 1 (1) | 0 (0)
HYPOTHYROIDISM (Endocrine disorders) | 0 (0) | 1 (1)
MULTINODULAR GOITER (Endocrine disorders) | 0 (0) | 1 (1)
BEGINNING MACULOPATHY OF THE LEFT EYE (Eye disorders) | 0 (0) | 1 (1)
BILATERAL GLAUCOMA (Eye disorders) | 1 (1) | 0 (0)
EARLY CATARACTS-BOTH EYES (Eye disorders) | 0 (0) | 1 (1)
IRRITATION LEFT EYE (Eye disorders) | 0 (0) | 1 (1)
LEFT EYE MACULAR EDEMA (Eye disorders) | 1 (1) | 0 (0)
MINIMAL DIABETIC RETINOPATHY (Eye disorders) | 0 (0) | 1 (1)
PROLIFERATIVE RETINOPATHY (Eye disorders) | 0 (0) | 1 (1)
WORSENED GLAUCOMA (Eye disorders) | 1 (1) | 0 (0)
WORSENING OF DEGENERATIVE MACULOPATHY (Eye disorders) | 1 (1) | 0 (0)
ABDOMINAL BLOATING (Gastrointestinal disorders) | 2 (3) | 0 (0)
ABDOMINAL PAIN (Gastrointestinal disorders) | 2 (2) | 2 (2)
BLACK STOOL (Gastrointestinal disorders) | 1 (1) | 0 (0)
COLON POLYPS (Gastrointestinal disorders) | 2 (2) | 0 (0)
DIARRHEA (Gastrointestinal disorders) | 4 (4) | 2 (2)
DIARRHEA (DUE TO METFORMIN) (Gastrointestinal disorders) | 0 (0) | 1 (1)
DIGESTIVE DISORDERS (Gastrointestinal disorders) | 1 (1) | 0 (0)
ENTEROCOLLITIS ACUTA (Gastrointestinal disorders) | 1 (1) | 0 (0)
FLATULENCE (Gastrointestinal disorders) | 1 (1) | 0 (0)
GASTRO-INTESTINAL SIDE EFFECTS OF METFORMIN (Gastrointestinal disorders) | 0 (0) | 1 (1)
GASTROESOPHAGEAL REFLUX (Gastrointestinal disorders) | 1 (1) | 1 (1)
GASTROESOPHAGEAL REFLUX DISEASE (Gastrointestinal disorders) | 1 (1) | 0 (0)
GI REFLUX (Gastrointestinal disorders) | 0 (0) | 1 (1)
INDIGESTION (Gastrointestinal disorders) | 1 (1) | 0 (0)
INTERMITTENT DIARRHEA (Gastrointestinal disorders) | 1 (1) | 1 (1)
INTERMITTENT NAUSEA (Gastrointestinal disorders) | 0 (0) | 1 (1)
LESIONS ON TONGUE, LIP, AND THROAT. (Gastrointestinal disorders) | 1 (1) | 0 (0)
MULTIPLE SMALL STOMACH ULCERS (Gastrointestinal disorders) | 0 (0) | 1 (1)
NAUSEA (Gastrointestinal disorders) | 3 (3) | 4 (4)
RECTAL BLEEDING (Gastrointestinal disorders) | 0 (0) | 1 (1)
STOMACH CRAMPS (Gastrointestinal disorders) | 0 (0) | 1 (1)
TEETH PAIN (Gastrointestinal disorders) | 0 (0) | 1 (1)
TOOTH PAIN (Gastrointestinal disorders) | 0 (0) | 1 (1)
VOMITING (Gastrointestinal disorders) | 3 (3) | 1 (1)
VOMITING EPISODE (Gastrointestinal disorders) | 1 (1) | 0 (0)
VOMITTING (Gastrointestinal disorders) | 0 (0) | 1 (1)
ABDOMINAL BRUISING FROM SENSOR INSERTION SITE (General disorders) | 1 (1) | 0 (0)
ANASARCA (General disorders) | 0 (0) | 1 (1)
ATYPICAL CHEST PAIN (General disorders) | 2 (2) | 0 (0)
BLEEDING (General disorders) | 0 (0) | 1 (1)
BLEEDING FOLLOWING SENSOR INSERTION (General disorders) | 0 (0) | 1 (1)
BLEEDING FROM INFUSION SITE (General disorders) | 2 (2) | 0 (0)
BLEEDING FROM INFUSION SITE UPON REMOVAL (General disorders) | 1 (1) | 0 (0)
CHEST PAIN (General disorders) | 3 (3) | 2 (3)
EDEMA - BILATERAL LEGS (General disorders) | 0 (0) | 1 (1)
EDEMA IN BOTH LEGS (General disorders) | 0 (0) | 1 (1)
FATIGUE (General disorders) | 1 (1) | 1 (1)
FEET SWELLING (General disorders) | 1 (1) | 0 (0)
FEVER (General disorders) | 1 (1) | 0 (0)
FLU LIKE SYMPTOMS (General disorders) | 1 (1) | 0 (0)
FLU LIKE SYMPTOMS AFTER RECEIVING FLU VACCINATION (General disorders) | 1 (1) | 0 (0)
HERNIA (General disorders) | 1 (2) | 0 (0)
INCREASE OF SWELLING IN BOTH FEET (General disorders) | 1 (1) | 0 (0)
INFLAMMATION LEFT GROIN (General disorders) | 0 (0) | 1 (1)
INFLAMMATORY NODULE (General disorders) | 1 (1) | 0 (0)
INFUSION SITE PAIN (General disorders) | 1 (1) | 0 (0)
INTOLERANCE TO METFORMIN (General disorders) | 2 (2) | 0 (0)
PAIN (General disorders) | 1 (1) | 1 (2)
PERIPHERAL EDEMA (General disorders) | 1 (1) | 0 (0)
RASH AT SITE OF INFUSION INSERTION (General disorders) | 1 (1) | 0 (0)
REDNESS AROUND IPRO INSERTION SITE. (General disorders) | 0 (0) | 1 (1)
SOLITARY BENIGN CYST (General disorders) | 0 (0) | 1 (1)
SWELLING IN FEET, BILATERAL (General disorders) | 1 (1) | 0 (0)
SWELLING OF BOTH FEET (General disorders) | 0 (0) | 1 (1)
THORACIC PAIN (General disorders) | 0 (0) | 1 (1)
CHOLELITHIASIS (Hepatobiliary disorders) | 0 (0) | 1 (1)
ENLARGED LIVER (Hepatobiliary disorders) | 0 (0) | 1 (1)
HEPATIC CIRROSIS (Hepatobiliary disorders) | 0 (0) | 1 (1)
ALLERGIC RESPONSE (Immune system disorders) | 1 (1) | 0 (0)
ABDOMINAL WALL ABSCESS (Infections and infestations) | 1 (1) | 0 (0)
ABSCESS - NECK (Infections and infestations) | 1 (1) | 0 (0)
ABSCESS RIGHT BUTTOCKS (Infections and infestations) | 1 (1) | 0 (0)
ACUTE BRONCHITIS (Infections and infestations) | 2 (2) | 2 (3)
ACUTE CYSTITIS (Infections and infestations) | 1 (1) | 0 (0)
ACUTE GASTRO-ENTERITIS (Infections and infestations) | 1 (1) | 1 (1)
ACUTE TONSILLITIS (Infections and infestations) | 0 (0) | 1 (1)
BLADDER INFECTION (Infections and infestations) | 1 (1) | 0 (0)
BRONCHITIS (Infections and infestations) | 4 (5) | 9 (11)
BRONCHITIS ACUTE (Infections and infestations) | 1 (1) | 0 (0)
CELLULITIS (Infections and infestations) | 2 (3) | 2 (2)
CELLULITIS - RIGHT FOOT (Infections and infestations) | 0 (0) | 1 (1)
CELLULITIS ON LEFT ABDOMEN (Infections and infestations) | 1 (2) | 0 (0)
CELLULITIS ON RIGHT ABDOMEN (Infections and infestations) | 1 (1) | 0 (0)
CELLULITIS ON RIGHT LOWER ABDOMEN (Infections and infestations) | 1 (1) | 0 (0)
CELLULITIS TO BOTH LEGS. (Infections and infestations) | 1 (1) | 0 (0)
CERATOCONJUNCTIVITIS EPIDEMIC (Infections and infestations) | 1 (1) | 0 (0)
CHEST INFECTION (Infections and infestations) | 0 (0) | 1 (1)
CHRONIC BRONCHITIS (Infections and infestations) | 1 (1) | 0 (0)
COLD (Infections and infestations) | 2 (2) | 3 (4)
COMMON COLD (Infections and infestations) | 7 (8) | 4 (4)
CONDYLOMA (Infections and infestations) | 0 (0) | 1 (1)
DENTAL ABSCESS (Infections and infestations) | 0 (0) | 3 (3)
DIVERTICULITIS (Infections and infestations) | 0 (0) | 1 (1)
EAR INFECTION (Infections and infestations) | 1 (1) | 0 (0)
ERYSIPELAS (Infections and infestations) | 1 (1) | 0 (0)
FLU (Infections and infestations) | 3 (3) | 3 (3)
FLU-LIKE SYNDROME (Infections and infestations) | 1 (1) | 0 (0)
FOLLICITIS (INFLAMED HAIR FOLLICLES) (Infections and infestations) | 1 (1) | 0 (0)
FOLLICULITIS (Infections and infestations) | 2 (2) | 0 (0)
FUNGAL RASH - BILATERAL BREASTS (Infections and infestations) | 1 (1) | 0 (0)
GASTRO ENTERITIS (Infections and infestations) | 0 (0) | 1 (1)
GASTROENTERITIS (Infections and infestations) | 2 (3) | 6 (6)
H. PYLORI INFECTION (Infections and infestations) | 0 (0) | 1 (1)
HERPES SIMPLEX (Infections and infestations) | 1 (1) | 0 (0)
INFECTED TOE ON LEFT FOOT (Infections and infestations) | 0 (0) | 1 (1)
INFECTION IN LEFT HIP (Infections and infestations) | 0 (0) | 1 (1)
INFECTION OF UPPER LIP (Infections and infestations) | 1 (1) | 0 (0)
INFECTION ON RIGHT LOWER LEG (Infections and infestations) | 0 (0) | 1 (1)
INTERMITTEND URINARY TRACT INFECTION (Infections and infestations) | 0 (0) | 1 (1)
INTESTINAL INFECTION (Infections and infestations) | 0 (0) | 1 (1)
KIDNEY INFECTION (Infections and infestations) | 0 (0) | 1 (1)
LEFT EAR INFECTION (Infections and infestations) | 0 (0) | 1 (1)
LOCAL INFECTION AROUND PUMP CATETER INSERTION SITE (Infections and infestations) | 1 (1) | 0 (0)
LOCAL SKIN INFECTION AT NEEDLE SITE INJECTION (Infections and infestations) | 1 (1) | 0 (0)
LOWER RESPIRATORY TRACT INFECTION (Infections and infestations) | 0 (0) | 1 (1)
MIDDLE EAR INFECTION (OTITIS MEDIA) LEFT (Infections and infestations) | 1 (1) | 0 (0)
NASOPHARYNGITIS (Infections and infestations) | 2 (2) | 0 (0)
ONYCHOMYCOSIS RIGHT BIG TOE (Infections and infestations) | 1 (1) | 0 (0)
ONYCHOMYCOSIS. (Infections and infestations) | 0 (0) | 1 (1)
OTITIS MEDIA LATERALIS DEXTRI (Infections and infestations) | 1 (1) | 0 (0)
PENILE INFECTION (Infections and infestations) | 1 (1) | 0 (0)
PHARYNGITIS (Infections and infestations) | 1 (1) | 1 (1)
PHARYNGITIS. (Infections and infestations) | 0 (0) | 1 (1)
PNEUMONIA (Infections and infestations) | 2 (2) | 2 (2)
PROBABLE VIRAL GASTROENTERITIS (Infections and infestations) | 0 (0) | 1 (1)
RECURRENT SKIN INFECTIONS AFTER REMOVAL OF INFUSION SET (Infections and infestations) | 1 (1) | 0 (0)
RECURRENT SKIN INFECTIONS(INFUSION SITE)EXACERBATION OF AE-4 (Infections and infestations) | 1 (1) | 0 (0)
RESPIRATORY INFECTION (Infections and infestations) | 1 (1) | 0 (0)
SCROTAL ABSCESS (Infections and infestations) | 0 (0) | 1 (1)
SHINGLES (Infections and infestations) | 1 (1) | 0 (0)
SINUS COLD (Infections and infestations) | 1 (1) | 1 (2)
SINUS INFECTION (Infections and infestations) | 0 (0) | 3 (3)
SINUSITIS (Infections and infestations) | 0 (0) | 4 (4)
SKIN ABSCESS (Infections and infestations) | 1 (1) | 0 (0)
SUBCUTANOUSE ABCESS (Infections and infestations) | 1 (1) | 0 (0)
SUPERFICIAL SKIN INFECTION (Infections and infestations) | 0 (0) | 1 (1)
TONSILITIS (Infections and infestations) | 1 (1) | 0 (0)
TONSILLITIS (Infections and infestations) | 1 (1) | 0 (0)
TOOTH ABSCESS (Infections and infestations) | 1 (1) | 0 (0)
TOOTH DECAY (Infections and infestations) | 0 (0) | 1 (1)
TOOTH INFECTION (Infections and infestations) | 0 (0) | 1 (1)
UPPER RESPIRATORY INFECTION (Infections and infestations) | 2 (2) | 0 (0)
UPPER RESPIRATORY TRACT INFECTION (Infections and infestations) | 9 (11) | 1 (1)
UPPER RESPIRATORY TRACT INFECTION. (Infections and infestations) | 0 (0) | 1 (1)
URINARY INFECTION (Infections and infestations) | 0 (0) | 1 (2)
URINARY TRACT INFECTION (Infections and infestations) | 6 (6) | 3 (3)
VAGINAL CANDIDIASIS (Infections and infestations) | 1 (1) | 0 (0)
WORSENING SKIN ABSCESS, UNDERARM, BILATERALLY (Infections and infestations) | 1 (1) | 0 (0)
YEAST INFECTION (Infections and infestations) | 1 (1) | 0 (0)
ANKLE SPRAIN-RIGHT (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
ANTERIOR WEDGE COMPRESION FRACTURE OF T12 VERTEBRA (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
BRUISED LEFT KNEE (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
BURN (Injury, poisoning and procedural complications) | 1 (1) | 1 (1)
BURN OF TOES OF FEET (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
CONTUSION TO BUTTOCK (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
CONTUSIONS (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
CONTUSIONS TO LEFT ELBOW (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
DRY BRUISING (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
FALL (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
FALL - ABRASIONS TO BOTH KNEES (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
FRACTURE OF FIFTH METATHARSAL BONE RIGHT (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
FRACTURED RIGHT MALLEOLUS (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
HEAD TRAUMA RIGHT TEMPORAL REGION (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
HEAT STROKE (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
INJURY RIGHT LOWER LEG (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
LEFT 2ND DIGIT INDEX FINGER PROXIMAL PHALANX SKIN REMOVED (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
LEFT MENISCUS TEAR (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
LEFT THUMB DISLOCATION (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
POISON IVY (SKIN REACTION) (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
POSTERIOR MUSCLE STRAIN BETWEEN SHOULDER BLADES (SCAPULAE). (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
RECCURENCE OF ACHILLES TENDON RUPTURE (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
RIGHT LATERAL EPICONDYLITIS (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
RIGHT SHOULDER INJURY (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
SECOND DEGREE BURN ON RIGHT FOREFOOT (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
SOFT TISSUE INJURY TO NECK AND SHOULDERS (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
SPRAINED ANKLE (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
SPRAINED LEFT KNEE (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
SUPERFICIAL WOUNDS (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
EXCESSIVE WEIGHT GAIN (Investigations) | 1 (1) | 0 (0)
FECAL OCCULT BLOOD TEST POSITIVE (Investigations) | 0 (0) | 1 (1)
INCREASE OF GGT (Investigations) | 0 (0) | 1 (1)
INCREASED LIVER ENZYMES (Investigations) | 0 (0) | 1 (1)
INCREASED PRESSURE BEHIND THE RIGHT EYE (Investigations) | 1 (1) | 0 (0)
DIABETIC FOOT (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
DIABETIC FOOT (LT- TOE 5) (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
DIABETIC FOOT, LEFT TOE 3. (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
DYSLIPIDEMIA (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
HYPERCALCEMIA (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
HYPERGLYCEMIA (Metabolism and nutrition disorders) | 4 (4) | 0 (0)
HYPERLIPIDEMIA (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
HYPOMAGNESEMIA (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
RECURRING HYPERGLICEMIA (481 MG/DL) (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
RIGHT FOOT POSSIBLE GOUT (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
SEVERE HYPOGLYCEMIA (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
TYPE 1 FHH (FAMILIAL HYPOCALCIURIC HYPERCALCEMIA) (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
ADHESIVE CAPSULITIS (FROZEN SHOULDER) LEFT ARM (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
BACK PAIN (Musculoskeletal and connective tissue disorders) | 2 (2) | 1 (1)
BAKERｴS CYST (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
BILATERAL LEG PAIN BELOW KNEES (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
BUTTOCK PAIN (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
CALCANEAL SPUR (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
CHRONIC LUMBAGO (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
COXITIS (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
DECREASED RANGE OF MOTION RIGHT ARM (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
DETERIORATION OF RIGHT SHOULDER PAIN (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
DIFFUSE MUSCLE AND SKELETAL PAIN (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
DORSALGIA (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
ELBOW PAIN (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
EXACERBATION OF BURSITIS RIGHT HIP (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
EXACERBATION OF BURSITIS TO LEFT HIP (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
GENERALIZED MYALGIA (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
GONARTHROSIS TOGETHER WITH KNEE-JOINT EFFUSION (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
HEEL PAIN (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
INCREASED NECK PAIN (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
INFRAPETELLAR BURSITIS (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
KNEE PAIN (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
KNEE STIFFNESS. (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
LEFT ELBOW PAIN (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
LEFT HIP PAIN (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
LEG PAIN (CRAMPING AND SPASMS) (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
LEGS PAIN (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
LESION ON RIGHT 1ST METATARSAL (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
LOW BACK PAIN (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
LOWER BACK PAIN (Musculoskeletal and connective tissue disorders) | 0 (0) | 2 (2)
LUMBAGO (Musculoskeletal and connective tissue disorders) | 2 (2) | 2 (2)
MUSCLE CRAMPS (Musculoskeletal and connective tissue disorders) | 0 (0) | 2 (2)
MUSCLE PAIN (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
NECK PAIN (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
PAIN IN THE HEEL BONE (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
PAIN LEFT ARM -EXACERBATION OF PREEXISTING CONDITION (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
PAIN LEFT SHOULDER (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
PAIN WITH HIS SHOULDER (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
POST TRAUMA LEFT HAND PAIN (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
PREPATELLAR BURSITIS (RIGHT KNEE) (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
RIGHT FLANK PAIN (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
RIGHT KNEE ARTHROSIS (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1)
RIGHT KNEE PAIN (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
RIGHT SHOULDER PAIN (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
RIGHT SIDED BACK PAIN (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
SEVERE BACK PAIN (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
SPINAL COLUMN ARTHROSIS (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
TENOSYNOVITIS OF THE RIGHT HAND-JOINT (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
TORTICOLIS (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
TRIGGER FINGER (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
VASOVAGAL EPISODE (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
WORSENING OF JOINTS PAIN (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
WORSENING OF PAIN LEFT LEG (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
WORSENING RIGHT SHOULDER PAIN (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
BASAL CELL CARCINOMA - RIGHT EAR (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
LESION(LIPOMA) OF SKIN (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
OSTEOCHONDROMA, RIGHT HALLUX (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
PLANTARS WART TO LEFT HEEL. (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
VERRUCAE VULGARIS (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
CARPAL TUNNEL SYNDROME (Nervous system disorders) | 0 (0) | 1 (1)
CARPEL TUNNEL SYNDROME (Nervous system disorders) | 0 (0) | 1 (1)
CEPHALALGIA (Nervous system disorders) | 1 (1) | 0 (0)
CERVICAL RADICULOPATHY ON C8 (Nervous system disorders) | 0 (0) | 1 (1)
DIZZINESS (Nervous system disorders) | 1 (1) | 3 (3)
ELECTIVE SURGERY FOR CARPAL TUNNEL SYNDROME ON LEFT HEND (Nervous system disorders) | 0 (0) | 1 (1)
EXACERBATION OF CARPEL TUNNEL SYNDROME (Nervous system disorders) | 1 (1) | 0 (0)
EXACERBATION OF PERIFERAL SENSORY NEUROPATHY (Nervous system disorders) | 0 (0) | 1 (1)
HEADACHE (Nervous system disorders) | 3 (3) | 3 (3)
INTERMITTENT DIZZINESS (Nervous system disorders) | 1 (1) | 0 (0)
INTERMITTENT NUMBNESS BOTTOM OF RIGHT FOOT (Nervous system disorders) | 0 (0) | 1 (1)
LOWER LIMBS NEUROPATHIC PAIN (Nervous system disorders) | 1 (1) | 0 (0)
NEUROPATHY (Nervous system disorders) | 1 (1) | 0 (0)
PARESTHESIA OF HANDS AND TOES (Nervous system disorders) | 0 (0) | 1 (1)
PARESTHESIAS IN BOTH FEET (Nervous system disorders) | 0 (0) | 1 (1)
POSTURAL DIZZINESS (Nervous system disorders) | 0 (0) | 1 (1)
RECURRENT HEADACHE (Nervous system disorders) | 1 (1) | 0 (0)
RECURRENT HEADACHES(INTERMITTENT) (Nervous system disorders) | 1 (1) | 0 (0)
SCIATIC (Nervous system disorders) | 0 (0) | 1 (1)
SCIATICA (Nervous system disorders) | 1 (1) | 0 (0)
SYNCOPE (Nervous system disorders) | 1 (1) | 0 (0)
TREMOR (Nervous system disorders) | 0 (0) | 1 (1)
VAGAL FAINTNESS (Nervous system disorders) | 1 (1) | 0 (0)
ANXIETY (Psychiatric disorders) | 1 (1) | 0 (0)
DEPRESSION (Psychiatric disorders) | 0 (0) | 2 (2)
EXACERBATION OF PRE EXISTING CONDITION-DEPRESSION (Psychiatric disorders) | 0 (0) | 1 (1)
EXACERBATION OF SYMPTOMS OF DEPRESSION (Psychiatric disorders) | 0 (0) | 1 (1)
INSOMNIA (Psychiatric disorders) | 0 (0) | 1 (1)
STRESS (Psychiatric disorders) | 1 (1) | 0 (0)
WORSENING ANXIETY (Psychiatric disorders) | 1 (1) | 0 (0)
WORSENING OF DEPRESSION (Psychiatric disorders) | 1 (1) | 1 (1)
BURNING SENSATION WITH MICTURITION (Renal and urinary disorders) | 1 (1) | 0 (0)
DIABETIC NEPHROPATHY (Renal and urinary disorders) | 1 (1) | 0 (0)
HEMATURIA (Renal and urinary disorders) | 0 (0) | 1 (1)
KIDNEY STONES (Renal and urinary disorders) | 0 (0) | 1 (1)
PROTEINURIA (Renal and urinary disorders) | 1 (1) | 0 (0)
RENAL COLIC (Renal and urinary disorders) | 0 (0) | 1 (1)
RENAL CYST (Renal and urinary disorders) | 1 (1) | 0 (0)
RENAL FUNCTION WORSENING. (Renal and urinary disorders) | 0 (0) | 1 (1)
BALANITIS PREPUTIAL (Reproductive system and breast disorders) | 0 (0) | 1 (1)
BENIGN HYPERTROPHY OF PROSTATA (Reproductive system and breast disorders) | 0 (0) | 1 (1)
BENIGN PROSTATE HYPERTROPHY (Reproductive system and breast disorders) | 1 (1) | 0 (0)
ENLARGED PROSTATE (Reproductive system and breast disorders) | 0 (0) | 1 (1)
ERECTILE DYSFONCTION (Reproductive system and breast disorders) | 0 (0) | 1 (1)
LEFT OVARIAN CYST (Reproductive system and breast disorders) | 1 (1) | 0 (0)
CHRONIC COUGH (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1)
DYSPNEA (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
EPISTAXIS (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
NASAL CONGESTION (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
NON PRODUCTIVE COUGH (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
PLEURISY (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
PLEURITIS (INFLAMMATION OF PLEURA) (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
PNEUMOPATHY (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
RESTRICTIVE LUNG DISEASE (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
SHORTNESS OF BREATH (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
SLEEP APNEA (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
SORE THROAT (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
UPPER RESPIRATORY TRACT INFLAMATION (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
0.5CM SKIN ULCER (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
2MM SCABBED ROUND LESION (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
ALLERGIC SKIN REACTION TO PLASTER(ADHESIVE OF INFUSION SET) (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
BLISTER ON BOTH FIRST METATARSALS (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
CONTACT DERMATITIS (BILATERAL HANDS) (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
DERMATITIS (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
ECCHYMOSIS (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
ECZEMA (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
ECZEMA ON LEFT EAR BACK (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
HIVES (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
INGROWN RIGHT HALLUX TOE NAIL LATERAL BORDER WITH PARONYCHIA (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
INGROWN TOENAIL (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
INGROWN TOENAIL SURGERY (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
LIPODYSTROPHY (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
LIPOHYPERTROPHY (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
MILD ALLERGIC REACTION TO ADHESIVE (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
PERIORBITAL OEDEMA (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
RED RASH ON ABDOMEN (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
SKIN LESION(BACK) (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
SKIN ALLERGIC REACTION TO ADHESIVE TAPE (OVERTAPE) (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
SKIN INFLAMMATION ON ABDOMEN (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
SKIN IRRITATION FROM INFUSION SITE ADHESIVE (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
SKIN LESION RIGHT 1ST PHALANGE PLANTAR ASPECT (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
SUBCUTANEOUS NODULE (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
RIGHT ROTATOR CUFF REPAIR (SURGERY) (Surgical and medical procedures) | 1 (1) | 0 (0)
VASECTOMY (Surgical and medical procedures) | 0 (0) | 1 (1)
WISDOM TOOTH EXTRACTION LEFT SIDE (Surgical and medical procedures) | 1 (1) | 0 (0)
DEEP VEIN THROMBOSIS - LEFT CALF (Vascular disorders) | 1 (1) | 0 (0)
HOT FLASH (Vascular disorders) | 1 (1) | 0 (0)
HYPERTENSION (Vascular disorders) | 4 (4) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days